CLINICAL TRIAL: NCT04262648
Title: Randomized, Blinded, Placebo-controlled, Study of Clinical and Laboratory Effects of L. Reuteri NCIMB 30351 in Functional Disorders of Gastrointestinal Tract and Skin Symptoms of Food Allergy in Children During the First Months of Life
Brief Title: Randomized Placebo-controlled Study of L. Reuteri NCIMB 30351 in GI Functional Disorders and Food Allergy in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoNatum Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioAmicus-001
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Infantile Colic; Constipation; Infantile Diarrhea; Gastro Esophageal Reflux
MeSH Terms: conditions — Colic; Constipation; Diarrhea, Infantile; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Dietary Supplement: Lactobacillus Reuteri
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri — Lactobacillus Reuteri NCIMB 30351
  Other Names: BioAmicus Lactobacillus drops
  Arms: Treatment
Dietary Supplement: Placebo — Sunflower oil
  Arms: Control

SUMMARY:
This study is a randomized, placebo-controlled, single-masked (blinded), post-marketing clinical study of a drug Lactobacillus Reuteri NCIMB 30351 drops in functional disorders of gastrointestinal tract and skin symptoms of food allergies in children between the ages of one and four months inclusive.

The aim of the study is to assess clinical effects of probiotics Lactobacillus Reuteri NCIMB 30351 drops on the symptoms of infantile colic, constipation, diarrhea, gastroesophageal reflux, atopic dermatitis/eczema in full-term newborns during the first months of life, laboratory parameters of microbiome will also be assessed.

A prospective study comparing two treatment groups:

Group 1 (treatment group) - 60 infants. Group 2 (control group) - 30 infants, placebo. The study drug will be taken in 1 time per day within 25 days. Allowed symptomatic therapy includes defoamers (simethicone-based preparations), carminative preparations (dill water (fennel)), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Parents / guardians speak Russian, understand the essence of study, are informed about the purpose of the study, understand their rights and signed informed consent form (ICF).
2. Vaginal delivery.
3. Full-term newborn.
4. Age at the time of the signing of informed consent form 1-4 months 28 days.
5. Breast- and formula-fed infants.
6. Colic , constipation , diarrhea, regurgitation (single symptom or combination of several symptoms).
7. Infant does not have other deviations in health, which would require the appointment of a specialized diet
8. Parents / guardians can and ready to regularly fill out the proposed diary form.

Exclusion Criteria:

1. Born by Cesarean section.
2. Premature newborn.
3. Congenital abnormalities or other clinical manifestations that may interfere with the study.
4. Lactase food supplements.
5. Other probiotic drugs, antibiotics, enteric antiseptics, antifungal and antiprotozoal drugs.

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change in the number of infantile colics | 25 days from the start of treatment
  Infantile colics are defined according to IV Rome criteria

SECONDARY OUTCOMES:
Change in the number of constipations | 25 days from the start of treatment
  Constipation is defined according to IV Rome criteria
Change in the number of diarrhea cases | 25 days from the start of treatment
  Diarrhea is defined according to IV Rome criteria
Change in the number of gastroesophageal reflux (posseting) cases | 25 days from the start of treatment
  Gastroesophageal reflux is defined according to IV Rome criteria
Presence of skin symptoms of food allergy | 25 days from the start of treatment
  Presence or absence of skin symptoms of food allergy will be assessed by investigator during general skin examination
Change in 16S RNA sequencing | 25 days from the start of treatment
  16S RNA in stool
Change in concentrations of stool carbohydrates | 25 days from the start of treatment
  Carbohydrates concentrations will be measured in stool filtrate
Change in concentrations in stool filtrate of volatile fatty acids | 25 days from the start of treatment
  Following volatile fatty acids concentrations will be assessed: acetic, propionic, butyric, valeric, caproic and their isomers

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Tyrsin, Study Director — NovoNatum CEO
Locations (2):
- Russia (2):
  - Children's City Clinical Hospital named after Bashlyaeva, Healthcare department of Moscow city, Moscow
  - Medical Center "St. Andrew's Hospitals - NEBOLIT", Moscow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tyrsin OY, Tyrsin DY, Nemenov DG, Ruzov AS, Odintsova VE, Koshechkin SI, D Amico L. Effect of Lactobacillus reuteri NCIMB 30351 drops on symptoms of infantile functional gastrointestinal disorders and gut microbiota in early infants: Results from a randomized, placebo-controlled clinical trial. Eur J Pediatr. 2024 May;183(5):2311-2324. doi: 10.1007/s00431-024-05473-y. Epub 2024 Mar 1. PMID 38427038